CLINICAL TRIAL: NCT06205290
Title: A Global Phase 3, Randomized, Open-label, Multi-center Trial Designed to Compare the Efficacy and Safety of Lisocabtagene Maraleucel vs Investigator's Choice Options (Idelalisib + Rituximab or Bendamustine + Rituximab) in Adult Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL), Whose Disease Has Failed Treatment With Both BTKi and BCL2i Targeted Therapies (A Double Class Exposed Population)
Brief Title: A Study to Compare the Efficacy and Safety of Lisocabtagene Maraleucel vs Investigator's Choice Options in Adult Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma, Whose Disease Has Failed Treatment With Both BTKi and BCL2i Therapies
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA082-1170
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Small Lymphocytic lymphoma; B cell malignancies; CD19+ B cell malignancies; Non-Hodgkin lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — idelalisib; Rituximab; Bendamustine Hydrochloride; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Liso-cel Monotherapy (Experimental)
  Interventions: Biological: Liso-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Arm B: Investigator's Choice (Active Comparator)
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Biological: Liso-cel — Specified dose on specified days
  Other Names: JCAR017; Breyanzi®; BMS-986387; lisocabtagene maraleucel
  Arms: Arm A: Liso-cel Monotherapy
Drug: Idelalisib — Specified dose on specified days
  Other Names: Zydelig®
  Arms: Arm B: Investigator's Choice
Drug: Rituximab — Specified dose on specified days
  Other Names: Rituxan®; Mabthera®; Riximyo®; Truxima®
  Arms: Arm B: Investigator's Choice
Drug: Bendamustine — Specified dose on specified days
  Other Names: Bendeka®; Treanda®; Belrapzo®
  Arms: Arm B: Investigator's Choice
Drug: Fludarabine — Specified dose on specified days
  Other Names: Fludara®; Bendarabin®
  Arms: Arm A: Liso-cel Monotherapy
Drug: Cyclophosphamide — Specified dose on specified days
  Other Names: Endoxan®; Cytoxan®
  Arms: Arm A: Liso-cel Monotherapy

SUMMARY:
The purpose of this study is to compare the efficacy and safety of liso-cel vs Investigator's Choice options (idelalisib + rituximab or bendamustine + rituximab) in adult participants with R/R CLL or SLL, whose disease has failed treatment with both BTKi and BCL2i targeted therapies.

ELIGIBILITY:
Inclusion Criteria

* Must have what doctors call measurable disease, which will be evaluated before each participant take part of the study.
* Must have received both a BTKi and a BCL2i treatment, and their disease must have come back or not responded to treatment, or they must not have been able to tolerate the side-effects of the BTKi and/or BCL2i treatment(s).
* Must also have an ECOG performance score of 0 or 1, which means they are able to carry out their normal daily activities without any problems.

Exclusion Criteria

* Heart problems.
* Bleeding disorders.
* Active cancer in their brain.
* Other reasons include:.

  i) Having certain treatments in the past.

ii) Having certain infections that are not under control.

iii) Having certain brain conditions.

- Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-16 (Estimated); Primary Completion 2031-10-13 (Estimated); Study Completion 2031-10-13 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per independent review committee (IRC) assessment | Up to 5 years from the last participant randomized

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years from the last participant randomized
Complete Response Rate (CRR) per IRC assessment | Up to 5 years from the last participant randomized
CRR per investigators' assessment | Up to 5 years from the last participant randomized
Complete response with incomplete bone marrow recovery (CRi) | Up to 5 years from the last participant randomized
Minimal residual disease (MRD)-negativity rate | Up to 5 years from the last participant randomized
Overall Response Rate (ORR) per IRC assessment | Up to 5 years from the last participant randomized
ORR per investigators' assessment | Up to 5 years from the last participant randomized
Duration of Response (DOR) per IRC assessment | Up to 5 years from the last participant randomized
Duration of Complete Response (DOCR) per IRC assessment | Up to 5 years from the last participant randomized
PFS per investigators' assessment | Up to 5 years from the last participant randomized
Progression post next line of treatment (PFS-2) | Up to 5 years from the last participant randomized
Number of participants with Adverse Events (AEs) | Up to 5 years from the last participant randomized
Number of participants with Adverse Events of Special Interest (AESIs) | Up to 5 years from the last participant randomized
Number of participants with laboratory abnormalities | Up to 5 years from the last participant randomized
Time from randomization to first confirmed clinically meaningful improvement from baseline in the European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC QLQ-C30) | Up to 5 years from the last participant randomized
  The following domains on the EORTC QLQ-C30 will be assessed:
  * Fatigue
  * Physical functioning
  * Role functioning
  * Cognitive functioning
  * Global health status/quality of life (GHS/QoL)
Time from randomization to first confirmed clinically meaningful improvement from baseline in the European Quality of Life Module Chronic Lymphocytic Leukemia 17 (EORTC QLQ-CLL17) | Up to 5 years from the last participant randomized
  The following domains on the EORTC QLQ-CLL17 will be assessed:
  * Symptom burden
  * Physical condition/fatigue
Mean changes from baseline in the following key health-related quality of life (HRQoL) domains: GHS/QoL | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-C30
Mean changes from baseline in the following key HRQoL domains: Fatigue | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-C30
Mean changes from baseline in the following key HRQoL domains: Physical functioning | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-C30
Mean changes from baseline in the following key HRQoL domains: Role functioning | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-C30
Mean changes from baseline in the following key HRQoL domains: Cognitive functioning | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-C30
Mean changes from baseline in the following key HRQoL domains: Symptom burden | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-CLL17
Mean changes from baseline in the following key HRQoL domains: Physical condition/fatigue | Up to 5 years from the last participant randomized
  As assessed by EORTC QLQ-CLL17

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (48):
- United States (16):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Local Institution - 0023, Duarte, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - Local Institution - 0120, Atlanta, Georgia
  - St. Luke's Mountain States Tumor Institute : Boise, Boise, Idaho
  - Local Institution - 0058, Iowa City, Iowa
  - Local Institution - 0048, Saint Matthews, Kentucky
  - Local Institution - 0101, Minneapolis, Minnesota
  - Local Institution - 0121, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - St. David's South Austin Medical Center, Austin, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Local Institution - 0068, Morgantown, West Virginia
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Austria (2):
  - Local Institution - 0094, Salzburg
  - Local Institution - 0093, Vienna
- Belgium (2):
  - Local Institution - 0113, Yvoir, Namur
  - Local Institution - 0112, Leuven, Vlaams-Brabant
- France (6):
  - Local Institution - 0038, Lyon, Auvergne-Rhône-Alpes
  - Local Institution - 0122, Rennes, Brittany Region
  - Local Institution - 0036, Montpellier, Languedoc-Roussillon
  - Local Institution - 0035, Clermont-Ferrand
  - Local Institution - 0037, Paris
  - Local Institution - 0034, Toulouse
- Germany (6):
  - Local Institution - 0084, Dresden, Saxony
  - Local Institution - 0081, Leipzig, Saxony
  - Local Institution - 0083, Kiel, Schleswig-Holstein
  - Local Institution - 0082, Cologne
  - Local Institution - 0079, Heidelberg
  - Local Institution - 0080, Ulm
- Italy (2):
  - Local Institution - 0091, Milan, Milano
  - Local Institution - 0088, Bologna
- Netherlands (2):
  - Local Institution - 0114, Amsterdam, North Holland
  - Local Institution - 0117, Groningen
- Local Institution - 0073, Oslo, Norway
- Spain (6):
  - Local Institution - 0104, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0105, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Local Institution - 0107, Santander, Cantabria
  - Local Institution - 0108, Madrid, Madrid, Comunidad de
  - Local Institution - 0106, Valencia, Valenciana, Comunitat
  - Local Institution - 0103, Salamanca
- Local Institution - 0071, Huddinge, Sweden
- United Kingdom (4):
  - Local Institution - 0115, London, London, City of
  - Local Institution - 0109, London, London, City of
  - Local Institution - 0111, Leeds
  - Local Institution - 0110, Oxford

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html